CLINICAL TRIAL: NCT00265265
Title: Phase 1, Double-Blind, Placebo-Controlled Multiple Dose Assessment of Potential Interactions Between Intravenous Cocaine and Atomoxetine
Brief Title: Assessment of Potential Interactions Between Intravenous Cocaine and Atomoxetine - 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-CPU-0010-1
Record Dates: First submitted 2005-12-13; First posted 2005-12-14 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-08

CONDITIONS: Cocaine-Related Disorders
Keywords: Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Atomoxetine Hydrochloride

INTERVENTIONS:
Drug: Atomoxetine

SUMMARY:
The purpose of this study is to assess potential interactions between intravenous (i.v.) cocaine and atomoxetine (Strattera) administered orally in four escalating doses.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years of age who are not seeking treatment at the time of the study
* Must be able to provide written informed consent
* Must be within 20 percent of ideal body weight and weigh at least 45 kg
* Must meet DSM0IV diagnostic criteria for cocaine abuse or dependence
* Must currently be using cocaine as confirmed by a positive BE
* If female and of child bearing potential, must agree to the use of birth control

Exclusion Criteria:

- please contact the site directly for more information

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16
Dates: Start 2005-08; Primary Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Safety
Cardiovascular responses

SECONDARY OUTCOMES:
Cocaine craving
pharmacokinetic assessment
Psychological Effects of Cocaine
Abuse Liability
Mood and personality assessments

CONTACTS AND LOCATIONS:
Overall Officials: Louis Cantilena, M.D., Principal Investigator — Uniformed Services University of Health Science
Locations (1):
- Uniformed Services University of Health Science, Bethesda, Maryland, United States

REFERENCES:
- [Result] Cantilena L, Kahn R, Duncan CC, Li SH, Anderson A, Elkashef A. Safety of atomoxetine in combination with intravenous cocaine in cocaine-experienced participants. J Addict Med. 2012 Dec;6(4):265-73. doi: 10.1097/ADM.0b013e31826b767f. PMID 22987022